CLINICAL TRIAL: NCT06719349
Title: Single-Level Lateral Lumbar Interbody Fusion in Author's Modification: Clinical and Radiographic Outcomes
Brief Title: Lumbar Discopathy Decompression with Lateral Interbody Fusion: Radiological and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: Podkarpackie Oncological Center (Other)
Responsible Party: Principal Investigator, Grzegorz Guzik, PhD, MD, Head of the Department of Orthopedics and Traumatology, Podkarpackie Oncological Center
Other Study IDs: 02-2024
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Spine Degeneration; Fusion of Spine (Disease)
Keywords: Spine; Decompression; Interbody Fusion; Diskectomy
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single level decompression and LLIF: Patients with single-segment L1-L4 spine discopathy treated with lumbar spine fusion modified by the authors were included in this study

SUMMARY:
The aim of the study was to introduce a single-segment lumbar spine decompression and fusion with intervertebral implants through modified by the authors lateral lumbar approach. Functional, surgical and radiographic outcomes was evaluated.

ELIGIBILITY:
Inclusion Criteria:

Single-segment L1-L4 spine discopathy.

Exclusion Criteria:

Any other spinal diseases. More than one level of discopathy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We retrospectively reviewed the medical data of patients who underwent single-level LIF from January to December 2021 at the Orthopaedic Oncology Department in Brzozów and the Trauma and Orthopaedic Department in Stalowa Wola.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
the quality of life | 3 months after the surgery
  the quality of life according to the EQ-VAS - Euro-Quality of Life Visual Analoque Score
the functional status - Karnofsky scale | 3 months after the surgery
  patients' neurological status, functional status according to the Karnofsky scale
the functional status Oswestry Disability Index | 3 months after the surgery
  patients' neurological status, functional status according to the ODI - Oswestry Disability Index
the intensity of pain | 3 months after the surgery
  the intensity of pain according to the VAS - Visual AnalogueScale score

SECONDARY OUTCOMES:
Radiographic Outcomes: The Cross-Sectional Area of the Spinal Canal | 3 months after the surgery
  Based on pre- and postoperative MRI/RTG the following aspects were assessed: The Cross-Sectional Area of the Spinal Canal, the width and depth of disc extrusion, and the width of the lateral recesses of the spinal canal, anterior disc height lumbar lordosis angle and lumbar segmental angle.
Radiographic Outcomes: The Height and Width of the Intervertebral Foramina | 3 months after the surgery
  Based on pre- and postoperative MRI/RTG the following aspects were assessed: The Height and Width of the Intervertebral Foramina
Radiographic Outcomes: lumbar segmental angle. | 3 months after the surgery
  Based on pre- and postoperative MRI/RTG the following aspects were assessed: lumbar segmental angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Subcarpatian Oncology Centre, Brzozów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
The medical records of the patients who participated in the study cannot be shared based on the protection of natural persons with regard to the processing of personal data according to the guidelines of the European Data Protection Board.

REFERENCES:
- [Background] Schizas C, Theumann N, Burn A, Tansey R, Wardlaw D, Smith FW, Kulik G. Qualitative grading of severity of lumbar spinal stenosis based on the morphology of the dural sac on magnetic resonance images. Spine (Phila Pa 1976). 2010 Oct 1;35(21):1919-24. doi: 10.1097/BRS.0b013e3181d359bd. PMID 20671589
- [Background] Lin GX, Akbary K, Kotheeranurak V, Quillo-Olvera J, Jo HJ, Yang XW, Mahatthanatrakul A, Kim JS. Clinical and Radiologic Outcomes of Direct Versus Indirect Decompression with Lumbar Interbody Fusion: A Matched-Pair Comparison Analysis. World Neurosurg. 2018 Nov;119:e898-e909. doi: 10.1016/j.wneu.2018.08.003. Epub 2018 Aug 10. PMID 30099187
- [Background] Ozgur BM, Aryan HE, Pimenta L, Taylor WR. Extreme Lateral Interbody Fusion (XLIF): a novel surgical technique for anterior lumbar interbody fusion. Spine J. 2006 Jul-Aug;6(4):435-43. doi: 10.1016/j.spinee.2005.08.012. PMID 16825052